CLINICAL TRIAL: NCT00837811
Title: An Open Label Extension Study of Multiple Subcutaneous Doses of LY2127399 in Patients With Rheumatoid Arthritis.
Brief Title: An Open Label Extension Study in Participants With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11768; H9B-MC-BCDI (Other: Eli Lilly and Company); CTRI/2009/091/000765 (Registry Identifier: India)
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Results first posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — tabalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2127399 (Experimental)
  Interventions: Biological: LY2127399

INTERVENTIONS:
Biological: LY2127399 — 60 milligrams [(mg) with potential for dose escalation to 120 mg] subcutaneously every 4 weeks for 48 weeks

SUMMARY:
To evaluate the safety and tolerability of LY2127399 administered as subcutaneous injections for 48 weeks in participants with Rheumatoid Arthritis

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Women must not be pregnant, breastfeeding or be at risk to become pregnant during study participation
* Have participated in either Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928)

Exclusion Criteria:

* Have had, during Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928), any safety event, [including having a recent, ongoing, or serious infection, a serious drug reaction, or any adverse event (AE) that caused discontinuation from treatment] that in the opinion of the investigator poses an unacceptable risk to participation in the study.
* Have received, during Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928), any drug not allowed by the study protocol including unapproved drugs, biologic disease-modifying anti-rheumatic drugs (DMARDs), or live vaccines.
* Enrollment in any other clinical trial involving off-label use of an investigational drug or device, or enrollment in any other type of medical research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern time (UCT/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (62):
- United States (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesa, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Desert, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riverside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Maria, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jupiter, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vero Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zephyrhills, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hickory, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleburg Heights, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orangeburg, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesquite, Texas
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elizabeth Vale, South Australia, Australia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège, Belgium
- Brazil (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campinas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Setor Oeste/Goiania
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitchener, Ontario
- Chile (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valdivia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viña del Mar
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hildesheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esztergom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kistarcsa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szolnok
- India (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lucknow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Secunderabad
- Mexico (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuernavaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampico
- Poland (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chełm Śląski
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş

REFERENCES:
- [Derived] Greenwald M, Szczepanski L, Kennedy A, Veenhuizen M, Komocsar WJ, Polasek E, Guerrettaz K, Berclaz PY, Lee C. A 52-week, open-label study evaluating the safety and efficacy of tabalumab, an anti-B-cell-activating factor monoclonal antibody, for rheumatoid arthritis. Arthritis Res Ther. 2014 Aug 29;16(4):415. doi: 10.1186/s13075-014-0415-2. PMID 25168268

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After ≥3 months treatment, investigator could choose 1-time dose increase [120 milligrams (mg) LY2127399 (LY)] for participants (pts) with ≥4 tender and ≥4 swollen joints. Additionally, 1-time dose decrease back to 60 mg LY permitted. Pts completing Week 72 completed study, but could be followed beyond Week 72 for B cell recovery (up to Week 112).
Groups:
- 60 mg LY2127399: LY2127399: 60 mg subcutaneous injections every 4 weeks for 48 weeks.
- 60/120 mg LY2127399: LY2127399: 60 mg subcutaneous injections every 4 weeks. After at least 3 months of treatment, participants had a dose increase to 120 mg LY2127399, administered once every 4 weeks. Participants remained at this dose level for the remainder of study treatment (48 weeks in total).
- 60/120/60 mg LY2127399: LY2127399: 60 mg subcutaneous injections every 4 weeks. After at least 3 months of treatment, the participant had a dose increase to 120 mg LY2127399, administered once every 4 weeks. Subsequently, the participant had a dose decrease back to 60 mg LY2127399, administered once every 4 weeks for the remainder of study treatment (48 weeks in total).
Period: Overall Study
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Started | 60 | 121 | 1
Received Any Amount of Study Drug | 60 | 121 | 1
Had at Least 1 Efficacy Assessment | 59 | 121 | 1
Included in Efficacy Analyses | 59 | 120 (Excludes participant from site with Good Clinical Practice (GCP) violations.) | 1
Completed | 53 | 87 | 0
Not Completed | 7 | 34 | 1
Not completed — Adverse Event | 4 | 6 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 11 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 9 | 0
Not completed — Sponsor Decision | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline was defined as Week 0 in this study [which is equivalent to Week 24 of the participant's prior study: Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928)]. The baseline characteristics of participants who received any amount of study drug and had at least 1 post-baseline efficacy assessment were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399 | Total
Number analyzed (Participants) | 59 | 121 | 1 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (11.86) | 51.5 (12.20) | 61.5 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable. | 52.2 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 99 | 1 | 150
  Male | 9 | 22 | 0 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 80 | 1 | 115
  Black or African American | 1 | 12 | 0 | 13
  Hispanic | 19 | 24 | 0 | 43
  East Asian | 5 | 4 | 0 | 9
  West Asian | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 3 | 3 | 0 | 6
  Australia | 1 | 0 | 0 | 1
  Belgium | 0 | 1 | 0 | 1
  Brazil | 4 | 9 | 0 | 13
  Canada | 0 | 4 | 0 | 4
  Chile | 5 | 8 | 0 | 13
  Germany | 1 | 1 | 0 | 2
  Hungary | 6 | 6 | 0 | 12
  India | 5 | 4 | 0 | 9
  Mexico | 12 | 12 | 0 | 24
  Poland | 12 | 30 | 0 | 42
  Puerto Rico | 0 | 1 | 0 | 1
  Romania | 3 | 3 | 0 | 6
  United States | 7 | 39 | 1 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE started on or after the date and time of the first dose of study drug administered in this study, or started prior to the study drug administration but worsened after the study drug started. Clinically significant events were defined as SAEs and other non-serious adverse events (AEs). A summary of SAEs and other non-serious AEs is located in the Reported Adverse Events module. Participants were on treatment up to 48 weeks. If a participant completed 48 weeks of treatment, the post-study treatment follow-up started at the next visit, 4 weeks later (Week 52). If a participant discontinued treatment early [early discontinuation (ED)], the post-study treatment follow-up started immediately afterwards. Baseline was defined as Week 0 in this study [which is equivalent to Week 24 of the participant's prior study: Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928)].
Time Frame: Baseline through Week 52 (up to 48 weeks of treatment or ED and follow-up through Week 52)
Population: Participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 60 | 121 | 1
Participants
  Any TEAE | 38 | 95 | 1
  Any SAE | 4 | 16 | 1

2. Primary Outcome: Number of Participants With Planned Laboratory Evaluations (Including Hematology, Clinical Chemistry, and Urinalysis) Reported as AEs
Description: For each planned laboratory evaluation, the range of values to be reported as AEs, regardless of causality, was pre-specified. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module. Baseline was defined as Week 0 in this study [which is equivalent to Week 24 of the participant's prior study: Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928)].
Time Frame: Baseline through Week 112
Population: Participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 60 mg LY2127399 Treatment: AEs reported while on study treatment (baseline up to Week 48) plus up to 3 weeks after discontinuation of study treatment (until next study visit).
  LY2127399: 60 mg subcutaneous injections every 4 weeks for 48 weeks.
- 60/120 mg LY2127399 Treatment: AEs reported while on study treatment (baseline up to Week 48) plus up to 3 weeks after discontinuation of study treatment (until next study visit).
  LY2127399: 60 mg subcutaneous injections every 4 weeks. After at least 3 months of treatment, participants had a dose increase to 120 mg LY2127399, administered once every 4 weeks. Participants remained at this dose level for the remainder of study treatment (48 weeks in total).
- 60/120/60 mg LY2127399 Treatment: AEs reported while on study treatment (baseline up to Week 48) plus up to 3 weeks after discontinuation of study treatment (until next study visit).
  LY2127399: 60 mg subcutaneous injections every 4 weeks. After at least 3 months of treatment, the participant had a dose increase to 120 mg LY2127399, administered once every 4 weeks. Subsequently, the participant had a dose decrease back to 60 mg LY2127399, administered once every 4 weeks for the remainder of study treatment (48 weeks in total).
- 60 mg LY2127399 Post-Study Treatment Follow-Up: AEs that started or worsened after discontinuation of study treatment (Week 52 or ED) through end of study (Week 72) plus 28 weeks, for participants who received only the 60 mg LY2127399 dose during study treatment.
  No study drug was administered during the post-study treatment follow-up.
- 60/120 mg LY2127399 Post-Study Treatment Follow-Up: AEs that started or worsened after discontinuation of study treatment (Week 52 or ED) through end of study (Week 72) plus 28 weeks, for participants who had a dose increase to 120 mg LY2127399 during study treatment.
  No study drug was administered during the post-study treatment follow-up.
- 60/120/60 mg LY2127399 Post-Study Treatment Follow-Up: AEs that started or worsened after discontinuation of study treatment (Week 52 or ED) through end of study (Week 72) plus 28 weeks, for participants who had a dose increase to 120 mg LY2127399 and subsequently, a dose decrease back to 60 mg LY2127399 during study treatment.
  No study drug was administered during the post-study treatment follow-up.
Arm/Group | 60 mg LY2127399 Treatment | 60/120 mg LY2127399 Treatment | 60/120/60 mg LY2127399 Treatment | 60 mg LY2127399 Post-Study Treatment Follow-Up | 60/120 mg LY2127399 Post-Study Treatment Follow-Up | 60/120/60 mg LY2127399 Post-Study Treatment Follow-Up
Number analyzed (Participants) | 60 | 121 | 1 | 60 | 121 | 1
Participants
  Alanine Aminotransferase (ALT) Increased | 0 | 1 | 0 | 0 | 1 | 0
  Aspartate Aminotransferase (AST) Increased | 0 | 1 | 0 | 0 | 1 | 0
  B-Lymphocyte Count Decreased | 0 | 0 | 0 | 0 | 1 | 0
  Blood Alkaline Phosphatase Increased | 0 | 1 | 0 | 0 | 0 | 0
  Blood Cholesterol Increased | 1 | 0 | 0 | 0 | 0 | 0
  Blood Immunoglobulin M (IgM) Increased | 0 | 0 | 0 | 0 | 1 | 0
  Gamma-Glutamyltransferase (GGT) Increased | 0 | 2 | 0 | 1 | 0 | 0
  Hepatic Enzyme Increased | 0 | 1 | 0 | 1 | 0 | 0
  Neutrophil Count Increased | 0 | 0 | 0 | 0 | 1 | 0
  Vitamin D Decreased | 1 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Count Increased | 0 | 0 | 0 | 0 | 1 | 0
  Dyslipidaemia | 0 | 1 | 0 | 0 | 0 | 0
  Hypercholesterolaemia | 0 | 2 | 1 | 0 | 0 | 0
  Hyperglycaemia | 0 | 1 | 0 | 0 | 0 | 0
  Hyperlipidaemia | 0 | 0 | 0 | 0 | 1 | 0
  Hypokalaemia | 0 | 0 | 1 | 0 | 1 | 0
  Vitamin B12 Deficiency | 0 | 1 | 0 | 0 | 0 | 0
  Vitamin D Deficiency | 0 | 0 | 0 | 0 | 1 | 0

3. Secondary Outcome: Change From Baseline in Tender Joint Count [Individual Component of the American College of Rheumatology (ACR) Core Set]
Description: The number of tender and painful joints was determined by examination of 28 joints (14 on each side) which included: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. Joints were assessed by pressure and joint manipulation on physical examination. The participant was asked for pain sensations on these manipulations and the investigator watched for spontaneous pain reactions. Any positive response on pressure, movement, or both was translated into a single tender-versus-nontender dichotomy. Baseline was defined as the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study. A decrease in tender joint count indicated an improvement in the participant's condition.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline tender joint assessment; excludes site with GCP issues; Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 59 | 120 | 1
tender joints | -9.2 (8.0) | -6.5 (8.2) | -12.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

4. Secondary Outcome: Change From Baseline in Swollen Joint Count (Individual Component of the ACR Core Set)
Description: The number of swollen joints was determined by examination of 28 joints (14 on each side) which included: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint. Baseline was defined as the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study. A decrease in swollen joint count indicated an improvement in the participant's condition.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline swollen joint assessment; excludes site with GCP issues; LOCF.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 59 | 120 | 1
swollen joints | -7.6 (6.8) | -5.3 (6.6) | 2.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

5. Secondary Outcome: Change From Baseline in Participant's Assessment of Disease Activity (Individual Component of the ACR Core Set)
Description: Participant's assessment of their current arthritis disease activity using a visual analog scale (VAS), which ranged from 0 millimeters (mm) (no arthritis activity) to 100 mm (extremely active arthritis). Baseline was defined as the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study. A decrease in disease activity score indicated an improvement in the participant's condition.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline self-rated assessment of disease activity; excludes site with GCP issues; LOCF.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 57 | 117 | 1
mm | -26.1 (27.1) | -16.7 (30.7) | -68.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

6. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity (Individual Component of the ACR Core Set)
Description: Physician's assessment of disease activity using a VAS that ranged from 0 mm (no arthritis activity) to 100 mm (extremely active arthritis). Baseline was defined as the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study. A decrease in disease activity score indicated an improvement in the participant's condition.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline physician's global assessment of disease activity; excludes site with GCP issues; LOCF.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 58 | 120 | 1
mm | -29.1 (23.6) | -18.4 (26.9) | -38.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

7. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index [(HAQ-DI) Individual Component of the ACR Core Set]
Description: The disability section of the health assessment questionnaire scored the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area, which ranged from 0 (no disability) to 3 (severe disability), were averaged to calculate HAQ-DI. Baseline was defined as the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study. A decrease in HAQ-DI score indicated an improvement in the participant's condition.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline HAQ-DI assessment; excludes site with GCP issues; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 59 | 118 | 1
units on a scale | -0.3 (0.5) | -0.3 (0.6) | -0.5 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

8. Secondary Outcome: Change From Baseline in Participant's Assessment of Joint Pain (Individual Component of the ACR Core Set)
Description: Participant's assessment of joint pain using a VAS, which ranged from 0 mm (no pain) to 100 mm (worst possible pain). Baseline was defined as the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study. A decrease in joint pain indicated an improvement in the participant's condition.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline self-rated assessment of joint pain; excludes site with GCP issues; LOCF.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 59 | 118 | 1
mm | -26.9 (26.4) | -13.4 (30.2) | -68.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

9. Secondary Outcome: Percent Change From Baseline in C-Reactive Protein [(CRP) Individual Component of the ACR Core Set]
Description: CRP is an indicator of inflammation. The percentage of change in CRP from baseline=[(post-baseline CRP-baseline CRP)/baseline CRP]*100. Baseline was defined as the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study. A negative change indicated an improvement in the participant's condition.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline CRP assessment; excludes site with GCP issues; LOCF.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 58 | 120 | 1
percent change | -11.1 (164.6) | 50.7 (214.4) | 241.4 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

10. Secondary Outcome: Percentage of Participants Achieving ACR20 Response
Description: ACR20 Responder Index: Composite of clinical, laboratory, and functional measures of rheumatoid arthritis. ACR20 Responder: had ≥20% improvement from baseline in both tender and swollen joint counts and ≥20% improvement in at least 3 of 5 criteria: participant's and physician's global assessment of disease activity, HAQ-DI (which measured participants' perceived degree of difficulty performing daily activities), joint pain, and CRP. Percentage of participants achieving ACR20 response=(number of ACR20 responders/number of participants treated)*100. Participants who discontinued from study prior to Week 52 were imputed as non-responders. Participants who reached Week 52 but had ≥1 of 7 components missing had missing components imputed by LOCF. This composite data imputation was denoted as non-responder imputation (NRI)/LOCF. Baseline: the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline ACR20 assessment; excludes site with GCP issues; missing data imputed by NRI/LOCF. Four (4), 29, and 1 participants were imputed as non-responders for the 60 mg, 60/120 mg, and 60/120/60 mg LY2127399 groups, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 59 | 120 | 1
percentage of participants | 66.1 [52.6 to 77.9] | 32.5 [24.2 to 41.7] | 0.0 [0.0 to 97.5]

11. Secondary Outcome: Percentage of Participants ACR50 Response
Description: ACR50 Responder Index: Composite of clinical, laboratory, and functional measures of rheumatoid arthritis. ACR50 Responder: had ≥50% improvement from baseline in both tender and swollen joint counts and ≥50% improvement in at least 3 of 5 criteria: participant's and physician's global assessment of disease activity, HAQ-DI (which measured participants' perceived degree of difficulty performing daily activities), joint pain, and CRP. Percentage of participants achieving ACR50 response=(number of ACR50 responders/number of participants treated)*100. Participants who discontinued from study prior to Week 52 were imputed as non-responders. Participants who reached Week 52 but had ≥1 of 7 components missing had missing components imputed by LOCF. This composite data imputation was denoted as NRI/LOCF. Baseline was defined as the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline ACR50 assessment; excludes site with GCP issues; missing data imputed by NRI/LOCF. Four (4), 29, and 1 participants were imputed as non-responders for the 60 mg, 60/120 mg, and 60/120/60 mg LY2127399 groups, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 59 | 120 | 1
percentage of participants | 33.9 | 13.3 | 0.0

12. Secondary Outcome: Percentage of Participants Achieving ACR70 Response
Description: ACR70 Responder Index: Composite of clinical, laboratory, and functional measures of rheumatoid arthritis. ACR70 Responder: had ≥70% improvement from baseline in both tender and swollen joint counts and ≥70% improvement in at least 3 of 5 criteria: participant's and physician's global assessment of disease activity, HAQ-DI (which measured participants' perceived degree of difficulty performing daily activities), joint pain, and CRP. Percentage of participants achieving ACR70 response=(number of ACR70 responders/number of participants treated)*100. Participants who discontinued from study prior to Week 52 were imputed as non-responders. Participants who reached Week 52 but had ≥1 of 7 components missing had missing components imputed by LOCF. This composite data imputation was denoted as NRI/LOCF. Baseline was defined as the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline ACR70 assessment; excludes site with GCP issues; missing data imputed by NRI/LOCF. Four (4), 29, and 1 participants were imputed as non-responders for the 60 mg, 60/120 mg, and 60/120/60 mg LY2127399 groups, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 59 | 120 | 1
percentage of participants | 18.6 | 6.7 | 0.0

13. Secondary Outcome: ACR-N Response
Description: The ACR-N Responder Index was a composite of clinical, laboratory, and functional measures of rheumatoid arthritis. This index was defined as the lowest of either a) percent change in tender joint count, b) percent change in swollen joint count, or c) median percent change in 5 core ACR criteria: participant global assessment of disease activity, physician global assessment of disease activity, HAQ-DI (which measured participants' perceived degree of difficulty performing daily activities), joint pain, and CRP. For example, a participant with an ACR-N of X had an improvement ≥X% in both tender and swollen joint counts and a median improvement ≥X% in the 5 criteria previously mentioned. Baseline was the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study. Results for the 60/120/60 mg LY2127399 treatment arm were not analyzed as the participant did not have an ACR assessment.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline ACR-N assessment; excludes site with GCP issues; LOCF. No participant was analyzed in the 60/120/60 mg LY2127399 treatment arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 59 | 120 | 0
units on a scale | 31.9 (47.6) | 11.3 (46.4) |

14. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Score
Description: The FACIT Fatigue Scale was a brief participant-reported measure of fatigue and consisted of 13 items. Scores ranged from 0 to 52, where higher scores indicated less fatigue. Baseline was defined as the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study. An increase in FACIT fatigue score indicated an improvement of the participant's condition.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline FACIT assessment; excludes site with GCP issues; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 59 | 118 | 1
units on a scale | 5.2 (10.4) | 5.1 (10.5) | -6.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

15. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28 Joint Count (DAS28)
Description: The DAS28 consisted of a composite score of the following variables: tender joint count (TJC28), swollen joint count (SJC28), CRP (milligrams per liter [mg/L]), and participant global assessment of his or her disease activity using a VAS (participant global VAS). The DAS28 was calculated by using the following formula: DAS28-CRP=0.56*square root(TJC28)+0.28*square root(SJC28)+0.36*natural log(CRP+1)+0.014*participant global VAS+0.96. Scores ranged from 1.0 to 9.4 where lower scores indicated less disease activity and remission is DAS28 <2.6. Baseline was defined as the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study. A decrease in DAS28 indicated an improvement in the participant's condition.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline DAS28 assessment; excludes site with GCP issues; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 56 | 117 | 1
units on a scale | -2.0 (1.5) | -1.3 (1.5) | -1.3 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

16. Secondary Outcome: Percentage of Participants With Response Based on European League Against Rheumatism Responder Index, 28 Joint Count (EULAR28)
Description: EULAR28 was defined by the participant's change from baseline in DAS28 score and the absolute DAS28 score achieved. DAS28 consisted of composite score of the following: tender joint count, swollen joint count, CRP, and participant global assessment of his\her disease activity (participant global VAS). EULAR28 categories included: No Response [improvement in DAS28 ≤0.6 units (u) or post-baseline DAS28 score >5.1 with improvement ≤1.2 u], Moderate Response (post-baseline DAS28 score ≤5.1 with improvement >0.6 u but <1.2 u or post-baseline DAS28 score >3.2 with improvement >1.2 u), and Good Response (post-baseline DAS28 score ≤3.2 with improvement >1.2 u). Baseline was the last assessment prior to the participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study. Percentage of participants=(number of participants with specific response/participants assessed)*100. Displayed percentages may not add up to 100% because of rounding.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline EULAR28 assessment; excludes site with GCP issues; LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 56 | 117 | 1
percentage of participants
  No response | 16.1 | 44.4 | 0
  Moderate response | 48.2 | 39.3 | 100.0
  Good response | 35.7 | 16.2 | 0

17. Secondary Outcome: Change From Baseline in Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) Component Scores
Description: SF-36 was a 36-item, health-related survey that assessed participant's quality of life on 8 domains: physical functioning, bodily pain, role limitations due to physical problems, role limitations due to emotional problems, general health, mental health, social functioning, vitality and 2 component scores (mental and physical health). Domain scores calculated by summing individual items for each domain and transforming scores into 0 to 100 scale; higher scores indicated better health status. The mental component summary (MCS) score, based on SF-36 domains, consisted of social functioning, vitality, mental health, and role-emotional scales (range: 0 to 100). The physical component summary (PCS) score, based on SF-36 domains, consisted of physical functioning, bodily pain, role-physical, and general health scales (range: 0 to 100). Baseline: last assessment prior to participant's first dose of LY2127399 in Study H9B-MC-BCDG (NCT00689728), Study H9B-MC-BCDH (NCT00785928), or this study.
Time Frame: Baseline, up to and through Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline SF-36 assessment; excludes site with GCP issues; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 59 | 117 | 1
units on a scale
  Physical Health Component Summary Score | 5.7 (8.0) | 4.1 (9.6) | 1.4 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.
  Mental Health Component Summary Score | 4.7 (12.2) | 2.9 (10.1) | -2.9 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

18. Secondary Outcome: Pharmacodynamics: Change From Baseline in Total B Cells [Cluster Designation 20+ (CD20+)] Absolute Cell Counts
Description: B-lymphocyte antigen CD20+ is an activated-glycosylated phosphoprotein expressed on the surface of all mature B cells. Baseline was defined as the last measurement prior to randomization to any treatment in either Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928). A negative change indicated a decrease in cell count.
Time Frame: Baseline, Weeks 52, 60, 72, 80, 88, and 100
Population: Participants who received any amount of study drug and a post-baseline total B cell assessment at the specified time points.
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/µL)
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 53 | 83 | 1
cells per microliter (cells/µL)
  Week 52: number analyzed (Participants) | 52 | 83 | 0
  Week 52 | -113.1 (103.4) | -110.3 (121.7) |
  Week 60: number analyzed (Participants) | 53 | 82 | 0
  Week 60 | -135.9 (119.0) | -143.1 (135.3) |
  Week 72: number analyzed (Participants) | 51 | 79 | 0
  Week 72 | -141.0 (105.4) | -151.6 (117.8) |
  Week 80: number analyzed (Participants) | 31 | 60 | 1
  Week 80 | -137.6 (85.7) | -150.9 (127.7) | -262.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.
  Week 88: number analyzed (Participants) | 22 | 45 | 1
  Week 88 | -109.9 (83.8) | -148.6 (131.3) | -143.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.
  Week 100: number analyzed (Participants) | 13 | 24 | 1
  Week 100 | -71.7 (68.7) | -127.3 (121.4) | -95.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

19. Secondary Outcome: Pharmacodynamics: Change From Baseline in Peripheral Blood B Cell Subsets (Absolute Cell Counts)
Description: Cell surface marker CD19, CD27, and immunoglobulin D (IgD) expression levels were used to define the various B cell subsets. Cell surface markers were defined as being either present (+) or absent (-). Peripheral blood B cell subsets included: mature naive cells (CD19+IgD+CD27-); immature/transitional cells (CD19+IgD-CD27-); switched memory (CD19+IgD-CD27+); and non-switched memory (CD19+IgD+CD27+). Baseline was defined as the last measurement prior to randomization to any treatment in either Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928). A negative change indicated a decrease in cell count.
Time Frame: Baseline, Weeks 52, 60, 72, 80, 88, and 100
Population: Participants who received any amount of study drug and had the specified peripheral blood B cell subset assessment post-baseline at the specified time points.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 52 | 82 | 1
cells/µL
  Mature Naive Cells, Week 52: number analyzed (Participants) | 52 | 82 | 0
  Mature Naive Cells, Week 52 | -115.0 (79.9) | -109.2 (92.2) |
  Mature Naive Cells, Week 60: number analyzed (Participants) | 4 | 0 | 0
  Mature Naive Cells, Week 60 | -138.8 (67.1) |  |
  Mature Naive Cells, Week 72: number analyzed (Participants) | 50 | 76 | 0
  Mature Naive Cells, Week 72 | -95.9 (75.4) | -102.6 (90.4) |
  Mature Naive Cells, Week 80: number analyzed (Participants) | 1 | 8 | 1
  Mature Naive Cells, Week 80 | -189.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable. | -80.1 (62.8) | -123.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.
  Mature Naive Cells, Week 88: number analyzed (Participants) | 2 | 6 | 0
  Mature Naive Cells, Week 88 | -116.5 (99.7) | -111.7 (75.5) |
  Mature Naive Cells, Week 100: number analyzed (Participants) | 0 | 2 | 0
  Mature Naive Cells, Week 100 |  | -89.0 (108.9) |
  Immature/Transitional Cells, Week 52: number analyzed (Participants) | 51 | 79 | 0
  Immature/Transitional Cells, Week 52 | -5.8 (7.10) | -4.5 (13.2) |
  Immature/Transitional Cells, Week 60: number analyzed (Participants) | 4 | 0 | 0
  Immature/Transitional Cells, Week 60 | -6.5 (7.9) |  |
  Immature/Transitional Cells, Week 72: number analyzed (Participants) | 50 | 74 | 0
  Immature/Transitional Cells, Week 72 | -8.6 (8.9) | -8.5 (15.5) |
  Immature/Transitional Cells, Week 80: number analyzed (Participants) | 1 | 7 | 1
  Immature/Transitional Cells, Week 80 | -5.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable. | -9.0 (12.1) | -10.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.
  Immature/Transitional Cells, Week 88: number analyzed (Participants) | 2 | 6 | 0
  Immature/Transitional Cells, Week 88 | -3.0 (4.2) | -9.0 (10.5) |
  Immature/Transitional Cells, Week 100: number analyzed (Participants) | 0 | 2 | 0
  Immature/Transitional Cells, Week 100 |  | -6.5 (0.7) |
  Switched Memory Cells, Week 52: number analyzed (Participants) | 52 | 82 | 0
  Switched Memory Cells, Week 52 | 12.6 (27.1) | 13.1 (31.4) |
  Switched Memory Cells, Week 60: number analyzed (Participants) | 4 | 0 | 0
  Switched Memory Cells, Week 60 | -6.5 (16.3) |  |
  Switched Memory Cells, Week 72: number analyzed (Participants) | 50 | 76 | 0
  Switched Memory Cells, Week 72 | -14.7 (18.9) | -17.7 (36.1) |
  Switched Memory Cells, Week 80: number analyzed (Participants) | 1 | 8 | 1
  Switched Memory Cells, Week 80 | -10.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable. | -7.5 (17.3) | -23.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.
  Switched Memory Cells, Week 88: number analyzed (Participants) | 2 | 6 | 0
  Switched Memory Cells, Week 88 | -10.0 (5.7) | -9.0 (10.2) |
  Switched Memory Cells, Week 100: number analyzed (Participants) | 0 | 2 | 0
  Switched Memory Cells, Week 100 |  | -13.0 (22.6) |
  Non-Switched Memory Cells, Week 52: number analyzed (Participants) | 51 | 79 | 0
  Non-Switched Memory Cells, Week 52 | 6.0 (22.0) | 8.3 (22.2) |
  Non-Switched Memory Cells, Week 60: number analyzed (Participants) | 4 | 0 | 0
  Non-Switched Memory Cells, Week 60 | -3.8 (2.2) |  |
  Non-Switched Memory Cells, Week 72: number analyzed (Participants) | 50 | 74 | 0
  Non-Switched Memory Cells, Week 72 | -10.5 (18.0) | -7.3 (18.7) |
  Non-Switched Memory Cells, Week 80: number analyzed (Participants) | 1 | 7 | 1
  Non-Switched Memory Cells, Week 80 | -4.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable. | -3.6 (4.3) | -35.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.
  Non-Switched Memory Cells, Week 88: number analyzed (Participants) | 2 | 6 | 0
  Non-Switched Memory Cells, Week 88 | -18.0 (17.0) | -8.2 (9.7) |
  Non-Switched Memory Cells, Week 100: number analyzed (Participants) | 0 | 2 | 0
  Non-Switched Memory Cells, Week 100 |  | -10.5 (9.2) |

20. Secondary Outcome: Pharmacodynamics: Change From Baseline in Serum Immunoglobulin
Description: Immunoglobulins, or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Change from baseline serum immunoglobulin G (IgG), immunoglobulin M (IgM), and immunoglobulin A (IgA) levels are reported. Baseline was defined as the last measurement prior to randomization to any treatment in either Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928). A negative change indicated a decrease in immunoglobulin levels.
Time Frame: Baseline, up to Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline serum immunoglobulin assessment; LOCF.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 59 | 121 | 1
grams per liter (g/L)
  IgG | -1.8 (2.1) | -2.0 (3.8) | -1.9 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.
  IgM | -0.3 (0.4) | -0.3 (0.5) | -0.2 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.
  IgA | -0.6 (0.8) | -0.5 (0.7) | -0.8 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

21. Other Pre Specified Outcome: Number of Participants Who Died, Any Cause
Description: A summary of serious and other non-serious AEs regardless of causality is located in the Reported Adverse Events module. Baseline was defined as Week 0 in this study [which is equivalent to Week 24 of the participant's prior study: Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928)]. Participants were on treatment up to 48 weeks. If a participant completed 48 weeks of treatment, the post-study treatment follow-up started at the next visit, 4 weeks later (Week 52). If a participant discontinued treatment early, the post-study treatment follow-up started immediately afterwards. After treatment discontinuation, participants could be followed beyond Week 72 for B cell recovery (up to Week 112).
Time Frame: Baseline through Week 52 (up to 48 weeks of treatment or ED and follow-up through Week 52) and post-study treatment follow-up (start of Week 53 or ED up to and through Week 72 and start of Week 73 up to and through Week 112)
Population: Participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 60 | 121 | 1
Participants
  Died on study treatment [up to Week (Wk) 52] | 0 | 1 | 0
  Died post-study treatment Wk 53/ED through Wk 72 | 1 | 0 | 0
  Died post-study treatment Wk 73 through Wk 100 | 1 | 1 | 0

22. Secondary Outcome: Pharmacodynamics: Change From Baseline in Rheumatoid Factor (RF) Levels at Week 52
Description: RF is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis. Higher RF levels indicate an aggressive rheumatoid arthritis and a higher risk of joint damage. Baseline was defined as Week 0 in this study [which is equivalent to Week 24 of the participant's prior study: Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928)]. A decrease in RF levels indicated an improvement in the participant's condition. Results for the 60/120/60 mg LY2127399 treatment arm were not analyzed as the participant did not have a Week 52 RF level assessment.
Time Frame: Baseline, Week 52
Population: Participants who received any amount of study drug and had Week 52 post-baseline RF level assessment, excluding the site with GCP issues. No participant was analyzed in the 60/120/60 mg LY2127399 treatment arm.
Measure: Mean (Standard Deviation); unit: international units/milliliter (IU/mL)
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399
Number analyzed (Participants) | 50 | 87
international units/milliliter (IU/mL) | -26.9 (241.4) | -53.8 (312.6)

23. Secondary Outcome: Pharmacodynamics: Change From Baseline in Serum Anti-Cyclic Citrullinated Peptide (Anti-CCP) Antibodies
Description: Anti-CCP antibodies were measured using an enzyme-linked immunosorbent assay (ELISA) method. In general, high levels of the antibody indicated an aggressive rheumatoid arthritis and a higher risk of joint damage. Baseline was defined as Week 0 in this study [which is equivalent to Week 24 of the participant's prior study: Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928)]. A decrease in anti-CCP antibodies indicated an improvement in the participant's condition.
Time Frame: Baseline, up to Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline anti-CCP assessment, excluding site with GCP issues; LOCF.
Measure: Mean (Standard Deviation); unit: units per milliliter (U/mL)
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 52 | 113 | 1
units per milliliter (U/mL) | 6.9 (241.9) | -19.4 (358.7) | 0.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

24. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assessed the rate at which red blood cells fell in a test tube. Normal range was considered to be 0 to 20 or 0 to 30 millimeters per hour (mm/h), depending on the reference range used by the laboratory. Higher scores indicated greater inflammation. Percent change from baseline ESR=[(post-baseline ESR- baseline ESR)/baseline ESR]*100. Baseline was defined as Week 0 in this study [which is equivalent to Week 24 of the participant's prior study: Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928)]. A decrease in ESR indicated an improvement in the participant's condition.
Time Frame: Baseline, up to Week 52
Population: Participants who received any amount of study drug and had at least 1 post-baseline ESR assessment, excluding site with GCP issues; LOCF.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 57 | 116 | 1
percent change | 5.0 (63.7) | 20.9 (103.9) | -25.0 (NA) — Only 1 participant in the analysis, therefore standard deviation is not calculable.

25. Secondary Outcome: Number of Participants With LY2127399 Immunogenicity (Anti-LY2127399 Antibodies)
Description: The number of participants who had treatment-emergent or follow-up emergent anti-LY2127399 antibodies [anti-drug antibodies (ADA)] is reported. Treatment-emergent was defined as participants who had any sample from baseline through Week 52 that was a 4-fold increase (2 dilution increase) in immunogenicity titer over the baseline titer, or participants who tested negative at baseline and positive post-baseline (at titer of ≥1:20). Follow-up emergent was defined as any sample during follow-up that was a 4-fold increase (2 dilution increase) in immunogenicity titer over the baseline titer. The number of participants with baseline positive ADA data is also reported. Baseline was defined as the last measurement prior to randomization to any treatment in either Study H9B-MC-BCDG (NCT00689728) or Study H9B-MC-BCDH (NCT00785928).
Time Frame: Baseline through Week 52 (up to 48 weeks of treatment or ED and follow-up through Week 52) and post-study treatment follow-up (start of Week 53 or ED up to and through Week 112)
Population: Participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg LY2127399 | 60/120 mg LY2127399 | 60/120/60 mg LY2127399
Number analyzed (Participants) | 60 | 121 | 1
Participants
  Baseline Positive ADA | 2 | 1 | 0
  Treatment-Emergent ADA | 6 | 15 | 0
  Follow-Up Emergent ADA: number analyzed (Participants) | 50 | 91 | 1
  Follow-Up Emergent ADA | 2 | 5 | 0

ADVERSE EVENTS:
Time Frame: Baseline through Week 52 (up to 48 weeks of treatment or ED and follow-up through Week 52) and post treatment follow-up (start of Week 53 or ED up to and through Week 112)
Description: Participants (pt) treated up to 48 weeks (wks). If pt completed 48 wks of treatment, post-study treatment follow-up started next visit, 4 wks later (Wk 52). If pt discontinued treatment early, post-study treatment follow-up started immediately afterwards. After treatment discontinuation, pts followed beyond Wk 72 for B cell recovery (up to Wk 112).
Groups:
- 60/120/60 mg LY2127399 Post-Study Treatment Follow-Up: AEs that started or worsened after discontinuation of study treatment (Week 52 or ED) through end of study (Week 72) plus 28 weeks, for participants who had a dose increase to 120 mg LY2127399 and a dose decrease back to 60 mg LY2127399 during study treatment.
  No study drug was administered during the post-study treatment follow-up.
Arm/Group | 60 mg LY2127399 Treatment | 60/120 mg LY2127399 Treatment | 60/120/60 mg LY2127399 Treatment | 60 mg LY2127399 Post-Study Treatment Follow-Up | 60/120 mg LY2127399 Post-Study Treatment Follow-Up | 60/120/60 mg LY2127399 Post-Study Treatment Follow-Up
Serious Adverse Events (participants affected / at risk) | 4/60 | 16/121 | 1/1 | 5/60 | 4/121 | 0/1
Other Adverse Events (participants affected / at risk) | 36/60 | 93/121 | 1/1 | 23/60 | 47/121 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 60 mg LY2127399 Treatment (N=60) | 60/120 mg LY2127399 Treatment (N=121) | 60/120/60 mg LY2127399 Treatment (N=1) | 60 mg LY2127399 Post-Study Treatment Follow-Up (N=60) | 60/120 mg LY2127399 Post-Study Treatment Follow-Up (N=121) | 60/120/60 mg LY2127399 Post-Study Treatment Follow-Up (N=1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTROPHIC CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEVICE DISLOCATION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS A (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA NECROTISING (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PSOAS ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRACHEAL OBSTRUCTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BENIGN LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OVARIAN EPITHELIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/51 (0) | 0/99 (0) | 0 (0) | 1/51 (1) | 0/99 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHEUMATOID LUNG (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTERIOSCLEROSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 60 mg LY2127399 Treatment (N=60) | 60/120 mg LY2127399 Treatment (N=121) | 60/120/60 mg LY2127399 Treatment (N=1) | 60 mg LY2127399 Post-Study Treatment Follow-Up (N=60) | 60/120 mg LY2127399 Post-Study Treatment Follow-Up (N=121) | 60/120/60 mg LY2127399 Post-Study Treatment Follow-Up (N=1)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPLINTER HAEMORRHAGES (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CERUMEN IMPACTION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EXTERNAL EAR INFLAMMATION (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPEN ANGLE GLAUCOMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ULCERATIVE KERATITIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL MUCOSAL ERUPTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SALIVARY GLAND ENLARGEMENT (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG INTOLERANCE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE HAEMORRHAGE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE NODULE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE PAIN (General disorders) | 2 (2) | 12 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE PARAESTHESIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE RASH (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHIOLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 6 (7) | 8 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HORDEOLUM (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTED BITES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
LABYRINTHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 5 (5) | 9 (9) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PHARYNGITIS (Infections and infestations) | 3 (3) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PHARYNGITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PHARYNGOTONSILLITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SIALOADENITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL PHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRACHEITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 12 (12) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 13 (13) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
VAGINAL ABSCESS (Infections and infestations) | 0/51 (0) | 0/99 (0) | 0 (0) | 0/51 (0) | 1/99 (1) | 0 (0)
VAGINAL INFECTION (Infections and infestations) | 0/51 (0) | 1/99 (1) | 0 (0) | 0/51 (0) | 0/99 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1/51 (1) | 1/99 (1) | 0 (0) | 0/51 (0) | 0/99 (0) | 0 (0)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRUG EXPOSURE DURING PREGNANCY (Injury, poisoning and procedural complications) | 0/51 (0) | 1/99 (1) | 0 (0) | 0/51 (0) | 0/99 (0) | 0 (0)
EPICONDYLITIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAIL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDON INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASPIRATION JOINT (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPIRATION PLEURAL CAVITY (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
B-LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD IMMUNOGLOBULIN M INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECG SIGNS OF VENTRICULAR HYPERTROPHY (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM ST SEGMENT ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEART RATE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
QRS AXIS ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITAMIN D DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WEIGHT INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATLANTOAXIAL INSTABILITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENTHESOPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FASCIITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOFASCIAL PAIN SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 10 (11) | 28 (30) | 0 (0) | 3 (3) | 14 (14) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BENIGN NEOPLASM OF THYROID GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADICULAR SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VASCULAR DEMENTIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITH NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROPATHY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 1/51 (1) | 0/99 (0) | 0 (0) | 0/51 (0) | 0/99 (0) | 0 (0)
METRORRHAGIA (Reproductive system and breast disorders) | 0/51 (0) | 0/99 (0) | 0 (0) | 1/51 (1) | 0/99 (0) | 0 (0)
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0/51 (0) | 1/99 (1) | 0 (0) | 0/51 (0) | 0/99 (0) | 0 (0)
UTERINE POLYP (Reproductive system and breast disorders) | 0/51 (0) | 1/99 (1) | 0 (0) | 0/51 (0) | 0/99 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0/51 (0) | 1/99 (1) | 0 (0) | 0/51 (0) | 0/99 (0) | 0 (0)
ALLERGIC COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYDROPNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RALES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECZEMA NUMMULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MACULE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN INDURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRODESIS (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CATARACT OPERATION (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEBRIDEMENT (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNOVECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH EXTRACTION (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AORTIC ARTERIOSCLEROSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 4 (4) | 8 (8) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHLEBITIS SUPERFICIAL (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENOUS INSUFFICIENCY (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Data integrity issues were identified at 1 study site involving 1 participant. Therefore, this site/participant is excluded from all efficacy analyses/results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days